CLINICAL TRIAL: NCT05213806
Title: The WHEAT International Trial: WithHolding Enteral Feeds Around Red Cell Transfusion to Prevent Necrotizing Enterocolitis in Preterm Neonates: an International, Multi-centre, Randomized Controlled Trial
Brief Title: WithHolding Enteral Feeds Around Blood Transfusion (International)
Acronym: WHEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Imperial College London (Other)
Responsible Party: Principal Investigator, Dr. Balpreet Singh, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1027137; 1025465 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2021-12-08; First posted 2022-01-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Necrotizing Enterocolitis
Keywords: Comparative Effectiveness Trial; Necrotizing Enterocolitis; Premature Infants; Blood Transfusion; Withholding enteral feeds
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Intervention Model Description: The WHEAT trial is a pragmatic, randomized, controlled, unblinded, international, multicentre, parallel-group superiority trial comparing two clinical care pathways.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Withholding feeds around transfusion (Active Comparator): All enteral feeds will be discontinued (the infant will be placed nil by mouth) for 4 hours prior to packed red cell transfusion, during the transfusion and until 4 hours post transfusion. During this period, hydration and blood glucose will be maintained according to local practice, commonly by providing parenteral nutrition or intravenous dextrose. Four hours after the red cell transfusion has finished, feeds will be recommenced to how they were being received prior to the decision to transfuse. This duration of withholding feeds will follow the approach used in other trials and observational studies, and identified as the most acceptable in a survey of UK neonatal units. It gives time for milk in the small bowel to transit into the large bowel before the transfusion and for the circulation to stabilize after the transfusion before milk feeds given into the stomach pass through into the small intestine.
  Interventions: Other: Withholding feeds around transfusion
- Continuing feeds around transfusion (Active Comparator): Enteral feeds will continue to be given prior, during and after the packed red cell transfusion, in the manner in which they were being given prior to the decision to transfuse. Infants will remain allocated to the same care pathway until 34(+6) weeks(+days) gestational age.
  Interventions: Other: Continued feeds around transfusion

INTERVENTIONS:
Other: Withholding feeds around transfusion — Withholding enteral feeds for preterm infants (<30 weeks) around the time of blood transfusions to determine if any impact on the development and/or severity of Necrotizing Enterocolitis.
  Arms: Withholding feeds around transfusion
Other: Continued feeds around transfusion — Continued enteral feeds
  Arms: Continuing feeds around transfusion

SUMMARY:
The WHEAT International trial is a comparative effectiveness trial exploring whether withholding enteral feeds around the time of blood transfusion in very premature infants (<30 weeks) will reduce the occurrence of Necrotizing Enterocolitis (NEC). Currently both continued feeding and withholding feeding are approved care practices. The current study will randomize infants from Neonatal Intensive Care Units (NICUs) across Canada and the United Kingdom (UK) into one of the two care approaches (withholding or continued feeds) to determine if any significant outcomes are found.

DETAILED DESCRIPTION:
BACKGROUND: Necrotizing enterocolitis (NEC) is a devastating disease that affects mostly the intestine of premature infants. The wall of the intestine is invaded by bacteria, which cause local infection and inflammation that can ultimately destroy the wall of the bowel (intestine). NEC is among the most potentially devastating neonatal diseases and has a mortality of up to 33%, the most severe form (requiring surgery or resulting in death) affects about 5% of infants born at less than 30 gestational weeks; survivors are at high risk of long-term health and developmental problems. Prevention of NEC has been identified as one of the most important research uncertainties in the field of preterm birth. A temporal association between red cell transfusion and the subsequent development of the disease is well described. This 'transfusion-associated NEC' may also be more severe with higher mortality. Very preterm or extremely low birth weight infants are among the most frequently transfused patients: between 56% and 90-95% have at least one transfusion, and those transfused received an average of 5 transfusions in their neonatal stay. Withholding milk feeds during red cell transfusion may reduce the risk of NEC by decreasing postprandial mesenteric ischemia but there may be harmful effects of pausing enteral feeds. However, due to a lack of good quality evidence, there is no consensus regarding the optimal feeding strategy during a blood transfusion.

Both comparator pathways of care are standard practice in Canada and the UK; the WHEAT trial is a comparative effectiveness trial. The two care pathways that will be compared are:

1. Withholding Feeds Around Transfusion: All enteral feeds will be discontinued (the infant will be placed nil by mouth) for 4 hours prior to packed red cell transfusion, during the packed red cell transfusion and until 4 hours post packed red cell transfusion.
2. Continuing Feeds Around Transfusion: Enteral feeds will continue to be given prior, during and after the packed red cell transfusion, in the manner in which they were being given prior to the decision to transfuse.

Infants will remain allocated to the same care pathway until 34(+6) weeks(+days) gestational age.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm birth at <30+0 gestational weeks + days

Exclusion Criteria:

1. Parent(s) opt-out of trial participation.
2. Packed red cell transfusion with concurrent enteral feeds prior to enrolment. (Infants who have received a packed red cell transfusion while nil-by-mouth are eligible; or minimal enteral nutrition (<15 ml/kg/day feeds) at the time of transfusion; defined as before, during and for at least 4 hours after transfusion, are eligible.
3. Infants who are not being fed at the time of randomization or where enteral feeding is contraindicated [e.g. Major congenital abnormality of the gastrointestinal tract (GIT)].
4. Previous episode of NEC Bell stage 2 or higher or SIP prior to first study packed cell transfusion.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4333 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
NEC Stage II | From randomization to 40 weeks postmenstrual age
  NEC stage II or more after the first transfusion (modified Bell staging criteria) - Clinical signs and symptoms plus pneumatosis or portal/hepatic air diagnosed by x-ray or other imaging techniques

SECONDARY OUTCOMES:
Severe NEC | From randomization to 40 weeks postmenstrual age
  Histologically or surgically confirmed or recorded on the death certificate. These infants will be identified as described in Battersby et al. which will include infants recorded as being transferred for surgery.
Death | From randomization to 40 weeks postmenstrual age
  All-cause mortality
Late onset sepsis | From randomization to 40 weeks postmenstrual age
  Culture positive sepsis, onset after 72 hours of life
Number of days with a central venous line in situ | From birth to date of discharge home
  Number of days with a central venous line in situ
Number of central line associated bloodstream infections | From randomization to 40 weeks postmenstrual age
  Includes laboratory-confirmed bloodstream infection and clinical sepsis
Duration of any parenteral nutrition in days | From birth to 40 weeks postmenstrual age
  Duration of any parenteral nutrition in days
Growth | At date of discharge home
  Weight and head circumference z score.
Spontaneous Intestinal Perforation | From randomization to 40 weeks postmenstrual age
  Histologically or surgically confirmed or recorded in the death certificate.
Duration of hospital stay | From birth to date of discharge home
  Total duration of neonatal care in days including all levels of care (intensive care, high dependency care, special care and ordinary care)
Bronchopulmonary Dysplasia (BPD)/Chronic Lung Disease | At 36 weeks postmenstrual age
  Requiring respiratory support at 36 weeks gestation
Retinopathy of prematurity (ROP) | From randomization to 40 weeks postmenstrual age
  ROP requiring treatment
Severe Brain Injury | At 40 weeks postmenstrual age
  Intraventricular haemorrhage (IVH) grade 3 or 4 or cystic periventricular leukomalacia (PVL)

CONTACTS AND LOCATIONS:
Overall Officials: Balpreet Singh, MD, Principal Investigator — IWK Health, Canada; Jon Dorling, MD, Principal Investigator — Princess Anne Hospital, UK; Chris Gale, MD, Principal Investigator — Imperial College London, UK
Locations (1):
- IWK Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battersby C, Longford N, Mandalia S, Costeloe K, Modi N; UK Neonatal Collaborative Necrotising Enterocolitis (UKNC-NEC) study group. Incidence and enteral feed antecedents of severe neonatal necrotising enterocolitis across neonatal networks in England, 2012-13: a whole-population surveillance study. Lancet Gastroenterol Hepatol. 2017 Jan;2(1):43-51. doi: 10.1016/S2468-1253(16)30117-0. Epub 2016 Nov 8. PMID 28404014
- [Background] Lopez-Reyes JC, Juarez-Campa M. [Integration of teaching, service and research in the health area]. Salud Publica Mex. 1988 Sep-Oct;30(5):714-28. No abstract available. Spanish. PMID 3217834
- [Background] Hintz SR, Kendrick DE, Stoll BJ, Vohr BR, Fanaroff AA, Donovan EF, Poole WK, Blakely ML, Wright L, Higgins R; NICHD Neonatal Research Network. Neurodevelopmental and growth outcomes of extremely low birth weight infants after necrotizing enterocolitis. Pediatrics. 2005 Mar;115(3):696-703. doi: 10.1542/peds.2004-0569. PMID 15741374
- [Background] Pankov GI, Zarubinskaia LG. [Participation of medical scientists in Don in the revolutionary movement]. Sov Zdravookhr. 1989;(6):61-2. No abstract available. Russian. PMID 2675329
- [Background] Duley L, Uhm S, Oliver S; Preterm Birth Priority Setting Partnership Steering Group. Top 15 UK research priorities for preterm birth. Lancet. 2014 Jun 14;383(9934):2041-2042. doi: 10.1016/S0140-6736(14)60989-2. No abstract available. PMID 24931684
- [Background] Seges RA, Kenny A, Bird GW, Wingham J, Baals H, Stauffer UG. Pediatric surgical patients with severe anaerobic infection: report of 16 T-antigen positive cases and possible hazards of blood transfusion. J Pediatr Surg. 1981 Dec;16(6):905-10. doi: 10.1016/s0022-3468(81)80844-5. PMID 6279816
- [Background] Stritzke AI, Smyth J, Synnes A, Lee SK, Shah PS. Transfusion-associated necrotising enterocolitis in neonates. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F10-4. doi: 10.1136/fetalneonatal-2011-301282. Epub 2012 Mar 23. PMID 22447991
- [Background] Blau J, Calo JM, Dozor D, Sutton M, Alpan G, La Gamma EF. Transfusion-related acute gut injury: necrotizing enterocolitis in very low birth weight neonates after packed red blood cell transfusion. J Pediatr. 2011 Mar;158(3):403-9. doi: 10.1016/j.jpeds.2010.09.015. Epub 2010 Nov 10. PMID 21067771
- [Background] Mally P, Golombek SG, Mishra R, Nigam S, Mohandas K, Depalhma H, LaGamma EF. Association of necrotizing enterocolitis with elective packed red blood cell transfusions in stable, growing, premature neonates. Am J Perinatol. 2006 Nov;23(8):451-8. doi: 10.1055/s-2006-951300. Epub 2006 Sep 28. PMID 17009195
- [Background] Cunningham KE, Okolo FC, Baker R, Mollen KP, Good M. Red blood cell transfusion in premature infants leads to worse necrotizing enterocolitis outcomes. J Surg Res. 2017 Jun 1;213:158-165. doi: 10.1016/j.jss.2017.02.029. Epub 2017 Feb 28. PMID 28601308
- [Background] Keir AK, Yang J, Harrison A, Pelausa E, Shah PS; Canadian Neonatal Network. Temporal changes in blood product usage in preterm neonates born at less than 30 weeks' gestation in Canada. Transfusion. 2015 Jun;55(6):1340-6. doi: 10.1111/trf.12998. Epub 2015 Feb 5. PMID 25652740
- [Background] Kirpalani H, Whyte RK, Andersen C, Asztalos EV, Heddle N, Blajchman MA, Peliowski A, Rios A, LaCorte M, Connelly R, Barrington K, Roberts RS. The Premature Infants in Need of Transfusion (PINT) study: a randomized, controlled trial of a restrictive (low) versus liberal (high) transfusion threshold for extremely low birth weight infants. J Pediatr. 2006 Sep;149(3):301-307. doi: 10.1016/j.jpeds.2006.05.011. PMID 16939737
- [Background] Jasani B, Rao S, Patole S. Withholding Feeds and Transfusion-Associated Necrotizing Enterocolitis in Preterm Infants: A Systematic Review. Adv Nutr. 2017 Sep 15;8(5):764-769. doi: 10.3945/an.117.015818. Print 2017 Sep. PMID 28916576
- [Background] Sahin S, Gozde Kanmaz Kutman H, Bozkurt O, Yavanoglu Atay F, Emre Canpolat F, Uras N, Suna Oguz S, Underwood MA. Effect of withholding feeds on transfusion-related acute gut injury in preterm infants: a pilot randomized controlled trial. J Matern Fetal Neonatal Med. 2020 Dec;33(24):4139-4144. doi: 10.1080/14767058.2019.1597844. Epub 2019 Mar 28. PMID 30890001
- [Background] Neu J. Necrotizing enterocolitis: the search for a unifying pathogenic theory leading to prevention. Pediatr Clin North Am. 1996 Apr;43(2):409-32. doi: 10.1016/s0031-3955(05)70413-2. PMID 8614608
- [Background] Battersby C, Longford N, Costeloe K, Modi N; UK Neonatal Collaborative Necrotising Enterocolitis Study Group. Development of a Gestational Age-Specific Case Definition for Neonatal Necrotizing Enterocolitis. JAMA Pediatr. 2017 Mar 1;171(3):256-263. doi: 10.1001/jamapediatrics.2016.3633. PMID 28046187